CLINICAL TRIAL: NCT00607568
Title: Atomoxetine Effects in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MIRECC HIC 0605001441; K02DA021304 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Physiological Stress
Keywords: physical stress; psychological stress
MeSH Terms: conditions — Stress, Psychological | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): atomoxetine 40mg per day
  Interventions: Drug: Atomoxetine
- 2 (Placebo Comparator): second arm is placebo, sugar pill
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — atomoxetine 40mg per day or placebo
  For Phase I, subjects will be assigned to atomoxetine or placebo for 4 days. Subjects will then have a 4-15 day washout period and will be crossed over to the alternative treatment for Phase II.

SUMMARY:
A total of 18 healthy volunteers will participate in this four-week, within-groups, double-blind, placebo-controlled study. The study has two phases separated by a 4 to 15-day washout period. Subjects will be randomly assigned to receive either 40 mg atomoxetine or placebo. For Phase I, subjects will be assigned to atomoxetine or placebo for 4 days. After receiving medication or placebo for three days, subjects will have a 6-hour laboratory session, where responses to physical and psychological stress of a 20 mg/70 kg (20 mg maximum) dose of d-amphetamine will be measured. Several physiological, hormonal, and subjective outcome measures will be obtained during the experimental sessions. Subjects will then have a 4-15 day washout period and will be crossed over to the alternative treatment for Phase II.

DETAILED DESCRIPTION:
This pilot study will examine the effects of a norepinephrine reuptake blocker, atomoxetine, on physiological and subjective responses to physical and psychological models of stress and oral amphetamine in healthy volunteers. The physical stress model will be the cold pressor test (CPT) and the psychological stress will be the paced auditory serial addition task (PASAT).

Our overall hypothesis is that atomoxetine treatment, compared to placebo, will attenuate the physiological and subjective responses to stress and d-amphetamine.

2. Research Design: Double-blind, placebo-controlled, within-groups, outpatient study.

3. Methodology: A total of 18 healthy volunteers will participate in this four-week, within-groups, double-blind, placebo-controlled study. The study has two phases separated by a 4 to 15-day washout period. Subjects will be randomly assigned to receive either 40 mg atomoxetine or placebo. For Phase I, subjects will be assigned to atomoxetine or placebo for 4 days. After receiving medication or placebo for three days, subjects will have a 6-hour laboratory session, where responses to physical and psychological stress of a 20 mg/70 kg (20 mg maximum) dose of d-amphetamine will be measured. Several physiological, hormonal, and subjective outcome measures will be obtained during the experimental sessions. Subjects will then have a 4-15 day washout period and will be crossed over to the alternative treatment for Phase II.

4. Findings: Since our last renewal, a total of 16 subjects signed the consent form. Among those, 6 subjects did not return after signing the consent form. An additional 2 subjects were randomized but did not complete the study. One subjects started 3 times was randomized 3 times therefore counted three times in enrollment. Currently still enrolling subjects. (2/7/07)

Have completed this study with 10 subjects, study was published. This study has been entered twice.

ELIGIBILITY:
Inclusion Criteria:

* Female and males age 18 yrs to 45 yrs
* Current history of good health and normal ECG
* not pregnant , nor breast feeding
* using acceptable birth control methods

Exclusion Criteria:

* History of heart disease, hypertension, renal or hepatic diseases, glaucoma,hyperthyroidism,
* Current use of psychotropic medication
* Current dependence on alcohol or on drugs or treatments for drug or alcohol addiction within the past 5 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Atomoxetine treatment, compared to placebo, will attenuate the physiological and subjective responses to stress and d-amphetamine | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University